CLINICAL TRIAL: NCT07040189
Title: Gustabor Phase 1 - AI-based Creation of a Nutritional Plan to Compensate for Chemotherapy-induced Taste Disorders
Acronym: GustaborPilot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: LMU Klinikum (Other); University Hospital Regensburg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Gustabor1
Record Dates: First submitted 2025-06-17; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma; GI Cancer; Taste Disorders
Keywords: taste disorders; AI
MeSH Terms: conditions — Multiple Myeloma; Gastrointestinal Neoplasms; Taste Disorders

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm, non-blinded intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm All patients within the study are included in the intervention arm (Experimental): Gustabor server - AI based web platform providing print-out of individual lifestyle tips and recipe recommendations based on the patient's individual data and taste disorder
  Interventions: Other: Gustabor server

INTERVENTIONS:
Other: Gustabor server — AI based web platform providing individual lifestyle tips and recipe recommendations based on the patient's individual data and taste disorder

SUMMARY:
The study investigates taste disorders that commonly occur during or after cancer treatment, often leading to issues such as malnutrition and treatment discontinuation. Although many non-pharmacological recommendations exist, it is unclear which methods are suitable for which individuals. This pilot study aims to use an AI-based, or rule-driven system to generate personalized recommendations based on patients' specific impairments and taste disorder. For the pilot study, the AI will be trained on recipes to create individualized meal plans, helping to identify foods that are likely to be better. The primary endpoint is the assessment of the nutritional intervention as helpful at the second visit within 12 weeks of inclusion.

DETAILED DESCRIPTION:
The primary goal of this pilot study is to evaluate the feasibility and perceived helpfulness of a web application using AI-supported, personalized dietary recommendations for patients experiencing taste disorders during or after cancer therapy. The primary endpoint is the assessment of the nutritional intervention as helpful at the second visit within 12 weeks of inclusion.

The study is a prospective, single-arm, non-blinded intervention study with a maximum duration of 12 weeks for individual participants. Participants will be identified on the ward or in outpatient centers during their clinical treatment routine. Study measures and progress assessments will also only take place during the chemotherapy administrations planned as part of the clinical treatment routine or during the follow-up visits.

Data is entered into the Gustabor portal together with study staff. Initially, anthropometric data, eating habits, taste experiences, and taste alterations are recorded via questionnaires. Taste thresholds for sweet, sour, salty, bitter, and umami are then assessed using taste strips. Based on these inputs, an AI system generates personalized recipe recommendations as well as recommendations for actions (e.g., cold meals recommended in case of metallic taste), which are printed and reviewed with the participant. Additionally, participants receive a flyer containing general dietary advice for oncology patients. At the start of the study and again after a period of at least three and up to twelve weeks (timed to fit clinical routines), the Patient-Generated Subjective Global Assessment (PG-SGA) score will be recorded, evaluating weight, symptoms, dietary intake, and physical activity. At the second visit it will be assessed which recommendations were implemented and how helpful they were perceived overall (primary endpoint) and in detail.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Suffering from one of the following tumor entities: Multiple myeloma or malignant tumor of the gastrointestinal tract
* Mainly oral nutrition
* Subjectively perceived tumor therapy-related taste disorder
* At least two clinical presentations planned within 12 weeks with a minimum interval of three weeks
* Ability to participate in nutritional intervention, including use of the online portal and implementation of recipe suggestions (e.g. resources and access to a kitchen), either independently or with third-party support (e.g. by relatives, outpatient care services).

Exclusion Criteria:

* Pregnancy
* Taste disorder explained by other causes (e.g. existing before therapy or COVID disease)
* Placement in an inpatient care facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient rating of the nutritional intervention as helpful | Within 12 weeks of inclusion
  Rating of the overall nutritional intervention as helpful at the second visit within 12 weeks after inclusion my means of questionnaire. Rating using a 3-point scale: "Tried it and it didn't help", "Was somewhat helpful" and "Was very helpful".

SECONDARY OUTCOMES:
Patient-generated Subjective Global Assessment (PG-SGA) Score | Within 12 weeks of inclusion
  PG-SGA measures four key areas: weight history, including recent unintentional weight loss; the presence of nutrition-impacting symptoms such as nausea, taste changes, and appetite loss; current food intake compared to normal levels; and functional status, which measures the ability to perform daily activities. Based on the responses, a numeric score is calculated, with higher scores indicating a greater risk of malnutrition and the need for dietary intervention.
Identification of measures that were perceived as helpful | Within 12 weeks of inclusion
  Feedback rating regarding the individual tested measures as helpful / not helpful.
  Rating using a 3-point scale: "Tried it and it didn't help", "Was somewhat helpful" and "Was very helpful".
Exploration of correlations between measures and taste perception, tumor type and ongoing tumor therapy | Within 12 weeks of inclusion
  Correlation of the 3-point rated individual measures with individual taste perceptions, tumor type and ongoing tumor therapy

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - LMU Klinikum, Munich, Bavaria
  - Universitätsklinikum Regensburg, Regensburg, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria